CLINICAL TRIAL: NCT01796262
Title: The Effects of DHA (DOCOSAHEXAENOIC ACID) on Attention Deficit and Hyperactivity Disorder
Brief Title: The Effects of DHA on Attention Deficit and Hyperactivity Disorder
Acronym: DADA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: DMF srl (Dietetic Metabolic Food) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EM-00-11
Record Dates: First submitted 2013-02-12; First posted 2013-02-21 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2015-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; DHA; neuropsychological task; fNIRS; Docosahexaenoic Acid; n-3 polyunsaturated fatty acid; cognition; behavior
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Behavior | interventions — Docosahexaenoic Acids; wheat germ oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wheat germ oil (Placebo Comparator): Wheat germ oil 250 mg pearl b.i.d. for six months
  Interventions: Dietary Supplement: Wheat germ oil
- docosahexaenoic acid (Active Comparator): DHA Richoil 250 mg pearl (DMF srl): b.i.d. for six months
  Interventions: Dietary Supplement: docosahexaenoic acid

INTERVENTIONS:
Dietary Supplement: docosahexaenoic acid — Supplementation with DHA Richoil 250mg pearl b.i.d. for six months
  Other Names: DHA Richoil (DMF srl)
  Arms: docosahexaenoic acid
Dietary Supplement: Wheat germ oil — Wheat germ oil 250 mg pearl b.i.d. for six months
  Other Names: Wheat germ oil 250 mg pearl
  Arms: Wheat germ oil

SUMMARY:
The purpose of this study is to determine whether docosahexaenoic acid (DHA) is effective in reducing Attention Deficit/Hyperactivity Disorder (ADHD) core symptoms in a clinical sample of children and adolescents with ADHD.

DETAILED DESCRIPTION:
The primary objective of this study is to investigate the relative efficacy and tolerability of omega-3 fatty acid supplementation, more specifically docosahexaenoic acid (DHA), in reducing attention-deficit/hyperactivity disorder (ADHD) symptoms in children. The present study is going to determine whether DHA supplementation induces modifications in fatty acid blood level and to evaluate the correlation between this possible modification and behavioral, neuropsychological and functional indexes. The study is a randomised, placebo-controlled double-blind intervention trial providing within- and between-group comparisons over 6 months. At the start of the study, the patients will be randomized to active treatment with DHA in a dose of one capsules twice daily, corresponding to a daily dose of 500 mg DHA, or to placebo (identical capsules with fishy odor containing 500 mg wheat germ oil). A total of 50 patients will be included in the study which is conducted in the Child Psychiatry Unit of "E. Medea" Scientific Institute (in northern Italy). The study participants are recruited from among patients assessed and diagnosed at this clinic, aged 6 to 14 years, who met DSM-IV criteria for a diagnosis of ADHD of any subtype (see Eligibility Criteria for further details). The study will also recruit 20 typically developing children to provide a control group at the start of the research for comparison of fatty acid blood level and other outcome measures (healthy children will not be included in the supplementation phase).

Clinical assessment will be made were made at three visits at the site: at baseline (Visit 1), 4 months (Visit 2) and 6 months (Visit 3). At Visits 1-2-3, a blood sample will be taken for analysis of the blood fatty acid profile. At Visit 1, informed consent is signed, inclusion and exclusion criteria are assessed, and the investigators make a medical evaluation, including medical and psychiatric history, assessment of diagnosis and comorbidity through parent interview according to DSM-IV criteria (DAWBA). A number of other examinations and instruments will be used, including height and weight, pulse and blood pressure, a neuromotor examination and an assessment of the general level of functioning with clinical scales and questionnaires completed by parents (see Outcome Measure Section for more details); several neuropsychological tests and reading test will be performed by a developmental neuropsychologist. At Visits 1-2, changes in the concentration of oxygenated Hb and deoxygenated Hb in prefrontal cortex during a computerized visual working memory task will be assessed in a subset of patients (10 children from each group) with functional Near-Infrared Spectroscopy. Visit 2 will included the same examinations and instruments as Visit 1, with the exception of the reading test; Visit 3 will included all the same measures as Visit 1, with the exception of the fNIRS. Parents will return every month at the clinic to assess the compliance (defined as taking the prescribed dosage on more than 70% of the days in the interval), to be interviewed about current medical symptoms and any adverse events or side effects, and to get the supplementation dosage for the following month.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ADHD based on DSM-IV criteria and confirmed with Development and Well-Being Assessment (DAWBA) interview
* Comorbid disorder accepted: mood disorder, anxiety disorder, oppositional defiant disorder, conduct disorder, learning disorder
* Total IQ equal or above 85
* Aged from 6 to 14 years

Exclusion Criteria:

* Autism, Schizophrenia or othe psychiatric disorder not included in inclusion criteria
* associated neurologic, genetic, infectious or metabolic disorder, or a seizure disorder
* present or past use of any psychoactive drugs

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2012-06; Primary Completion 2015-02 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in ADHD RS-IV total score | Baseline, month 4, and month 6
  ADHD rating scale IV Parent Version-Investigator completed

SECONDARY OUTCOMES:
Change in CPRS-R | Baseline, month 4, and month 6
  Conners Parent Rating Scale Revised
Change in CGI-S | Baseline, month 4, and month 6
  Clinical Global Impression - Severity
Change in C-GAS | Baseline, month 4, and month 6
  Children Global Assessment Scale
Change in CHQ | Baseline, month 4, and month 6
  Child Health Questionnaire Total Score
Change SDQ Total Score | Baseline, month 4, and month 6
  Strenght and Difficulties Questionnaires

OTHER OUTCOMES:
Change in Functional Neuroimaging (functional Near-Infrared Spectroscopy) | Baseline and month 4
  Changes in the concentration of oxygenated Hb and deoxygenated Hb in prefrontal cortex during a computerized visual working memory task
Change in Cognitive Measure (ANT) | Baseline, month 4, and month 6
  Amsterdam Neuropsychological Task
Change in Fatty Acid blood level | Baseline, month 4, and month 6
  Fatty Acid blood level

CONTACTS AND LOCATIONS:
Overall Officials: Maria Nobile, MD, PhD, Principal Investigator — IRCCS 'Eugenio Medea'
Locations (1):
- IRCCS Eugenio Medea, Bosisio Parini, Lecco, Italy

REFERENCES:
- [Derived] Gillies D, Leach MJ, Perez Algorta G. Polyunsaturated fatty acids (PUFA) for attention deficit hyperactivity disorder (ADHD) in children and adolescents. Cochrane Database Syst Rev. 2023 Apr 14;4(4):CD007986. doi: 10.1002/14651858.CD007986.pub3. PMID 37058600
- [Derived] Crippa A, Tesei A, Sangiorgio F, Salandi A, Trabattoni S, Grazioli S, Agostoni C, Molteni M, Nobile M. Behavioral and cognitive effects of docosahexaenoic acid in drug-naive children with attention-deficit/hyperactivity disorder: a randomized, placebo-controlled clinical trial. Eur Child Adolesc Psychiatry. 2019 Apr;28(4):571-583. doi: 10.1007/s00787-018-1223-z. Epub 2018 Sep 24. PMID 30246216
- [Derived] Crippa A, Agostoni C, Mauri M, Molteni M, Nobile M. Polyunsaturated Fatty Acids Are Associated With Behavior But Not With Cognition in Children With and Without ADHD: An Italian study. J Atten Disord. 2018 Aug;22(10):971-983. doi: 10.1177/1087054716629215. Epub 2016 Feb 9. PMID 26861157